CLINICAL TRIAL: NCT04676438
Title: Incidence and Risk Factors of Chronic (Persistant) Post-surgical Pain in Oncological Breast Surgery : a Prospective Cohort Study in a National Institute of Oncology
Brief Title: Persistant Post-mastectomy Pain in Breast Cancer : Incidence and Risk Factors
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Principal Investigator, Amine Souadka, Principal Investigator, Moroccan Society of Surgery
Other Study IDs: PPMP_INO
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Neoplasms; Pain, Postoperative; Pain, Chronic
Keywords: Breast Neoplasms; Pain, Postoperative; Mastectomy and pain syndrome
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain; Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving surgery breast surgery for cancer at National Institute of Oncology: No intervention will be administered

SUMMARY:
Post Mastectomy Pain Syndrome (PMPS) is a major complication of breast surgery responsible for depression and disability.

The project consists of a prospective cohort on patients going for oncological breast surgery at National Institute of Oncology of Rabat.

Chronic postoperative pain (CPP) remains a disturbing and obscure clinical problem, which could last for more than 3 months after surgery. The aim of present study was to assess the prevalence of CPP, investigate its impact on life quality and explore its potential risk factors. After informed consent was signed, patients receiving surgery under general anesthesia in Peking Union Medical College Hospital and other medical centers participating in this study during 2018 will be included. Patients' preoperative information will be collected from medical record, including basic demographic data, primary disease and previous chronic diseases. Intraoperative information will be obtained from anesthesia record, including surgical scope, duration, length and location of incisions and blood loss. Acute pain will be evaluated in the ward of the department of surgery, when an app will be installed on patients' mobile phones. Our long-term postoperative follow-up would be performed by sending out survey questionnaires via this app in the 4th, 8th, 16th, 32th, and 48th weeks after surgery. The survey covers questions regarding the intensity, characteristic, location and impact on daily activities of CPP. Information regarding treatment of CPP will also be collected, if any. All the data gained will be summarized in our database and analyzed.

DETAILED DESCRIPTION:
Type of work: This is an observational, prospective, open, data-driven, single-center study at the National Institute of Oncology (NIO) - Mohamed Ben Abdellah Hospital in Rabat, affiliated to Mohammed V University in Rabat.

The objective of the study we are proposing is to determine the incidence and risk factors of chronic post-surgical pain in oncological breast surgery on the Moroccan population operated on and followed at the Sheikha Fatma Center of the National Institute of 'Oncology of Rabat.

The main objective of the study is to:

- Determine the incidence of chronic post-surgical pain in carcinological breast surgery

The secondary objectives are:

* Determine the clinical characteristics of chronic post-surgical pain and in particular the proportion of neuropathic pain and / or post-mastectomy pain syndromes
* Identify the preoperative, intraoperative and postoperative risk factors of developing chronic post-surgical pain in the Moroccan population
* Determine the incidence of acute severe postoperative pain
* Determine the characteristics of acute postoperative pain
* Identify the risk factors for severe acute postoperative pain

Work flow:

* The medical care of patients will be free to the responsible practitioners, according to the usual practice
* Nursing staff will be informed of the study
* An investigator will be appointed after training in the protocol. He will be independent and not responsible for the nursing activity
* Patients eligible for the study will be identified during the pre-anesthetic consultation, carried out in the week before surgery
* The recorded agreements will be obtained during these consultations
* Patients will be included once admitted to the operating room and operated
* The data collected is presented in the observation book in the appendix with the definitions of the events and the entry rules
* The patients will be followed up and reviewed at 3 months and 6 months in surgery consultation for reassessment and completion of the observation book

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to sign an informed consent document
* More than 18 years of age
* All American Society of Anesthesiology classes
* Patient undergo for breast surgery

Exclusion Criteria:

* Patients who expressed their refusal to participate in the study
* Patients unable to express their non-opposition to participating in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergo breast surgery at National Institute of Oncology (Sheikha Fatma center)
Sampling Method: Probability Sample
Enrollment: 722 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Post-mastectomy pain | preoperative-3months postoperative
  Assessed via breast pain questionnaire, including severity, frequency, related symptoms, and functional impairment

CONTACTS AND LOCATIONS:
Overall Officials: Abdelilah Ghannam, MD, Principal Investigator — Mohammed V University in Rabat
Locations (2):
- Morocco (2):
  - National Institute of Oncology of Rabat, Rabat
  - National Institut of Oncology, Surgical oncology department, Rabat

IPD SHARING:
Plan to Share IPD: Undecided